CLINICAL TRIAL: NCT03307135
Title: Medical Spastic Patient Machine Interface MSPMI : Biomechanical and Electrophysiological Assessment of the Triceps Surae Spasticity
Acronym: MSPMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Compiègne University of Technology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC17_0028
Record Dates: First submitted 2017-08-29; First posted 2017-10-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Spasticity, Muscle
Keywords: Spasticity; electrophysiology; biomechanics; objective assessment
MeSH Terms: conditions — Muscle Spasticity | interventions — Physical Examination; Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simple Assessment group (Experimental): Intervention is a single evaluation with the MSPMI by two evaluators.
  Interventions: Device: single assessment with the MSPMI
- Hospitalization group (Experimental): Evaluation with the MSPMI by two evaluators on two consultations separate by a 7 days interval.
  Interventions: Device: double assessment with the MSPMI with 7 days of interval
- Treatment group (Experimental): Evaluation with the MSPMI by two evaluators before and after specific therapies proposed on our usual practices (Selective tibial neurotomy, anesthetic block or botulinum toxin intramuscular injection).
  Interventions: Device: double assessment with the MSPMI before and after treatment

INTERVENTIONS:
Device: single assessment with the MSPMI — Manually applied stretch with the MSPMI installed on the foot and shank at 3 different velocities on 2 positions (knee flexed and extended)
  Arms: Simple Assessment group
Device: double assessment with the MSPMI with 7 days of interval — Manually applied stretch with the MSPMI installed on the foot and shank at 3 different velocities on 2 positions (knee flexed and extended)
  Arms: Hospitalization group
Device: double assessment with the MSPMI before and after treatment — Manually applied stretch with the MSPMI installed on the foot and shank at 3 different velocities on 2 positions (knee flexed and extended)
  Arms: Treatment group

SUMMARY:
Spasticity is a disorder of the muscular tonus that occurs in disease including the upper motor neuron (strokes, spinal cord injuries, multiple sclerosis, traumatic brain injuries or cerebral palsies). It begins few hours after the neural aggression and last until the grave.

The most accepted definition refers to a velocity-dependent increase in stretch reflexes elicited by passive stretch (Lance definition) but new approaches prefers to distinguish neural (reflex) and non-neural (soft tissues alterations) components of the increase resistance to a passive stretch. This deficiency is a major cause of complications as walking impairment, pain or bone deformities and may require intensive therapies (intrathecal baclofen infusion, intramuscular toxin botulinium injection, surgery, etc). Despite its high frequency and the potential complications, only clinical scales (modified Ashworth scale and modified Tardieu scale essentially) with criticized metrological properties are available for daily assessment. The SPASM Consortium has published on 2005 recommendations for developing devices using both mechanical and electrophysiological parameters. The principle challenge was to ally parameters accuracy and utilization facility allowing quickly evaluation to the patient's bed. Few research team works on this topic but mostly on specific population and nowadays, no device has really crossed the door of laboratories.

This kind of tool would help us to improve the quality of the follow-up and to guide us between the choices of specific therapies.

The MSPMI has been created following these recommendations in the University of Technology of Compiègne, thanks to the collaboration between researchers of the UMR 7338 CNRS and a brain surgeon of the Nantes University Hospital. The patent was obtained on 2012. This device allows the assessment of the ankle plantar extensor (triceps surae) during a manually applied stretch movement. This muscle was selected as it is frequently involved and treated for spasticity.

This study aims to evaluate the metrological properties of the MSPMI (reliabilities, responsiveness, known group validity, construct validity, measurement errors and internal consistency) among a large cohort of patients with no restriction of etiologies recruited in the Nantes University Hospital.

DETAILED DESCRIPTION:
Evaluation will include medical histories and specific information about spasticity management and consequences. The patient will be assessed by two evaluators with the MSPMI installed on the foot and the shank. MSPMI allows the record of angular movement of the ankle (position, speed and acceleration), of biomechanics (stiffness, torque, work and power) and electromyography (root mean squared and integrated electromyography signals) of two chiefs of the triceps surae (medial gastrocnemius and soleus). Electromyography data will be recorded on a maximum voluntary contraction when the deficiency will permit it. After that, data will be recorded at 3 velocities (with respect to the clinical scale recommendations) on two different positions (knee flexed and extended), according to our clinical practice. The evaluation on day 0 will allow the assessment of inter-rater intra-session reproductibility, internal consistency, construct validity, measurement error and known group validity. If the patient is hospitalized, he will be included on the "hospitalization group" and a second evaluation following the same protocol will be done 7 days later (assessment of inter and intra-rater inter-session reproductibility). If a specific therapy (selective tibial neurotomy, anesthetic block or botulinum toxin intramuscular injection) is proposed, the patient will be included on the "treatment group" and a new evaluation will be done after the therapy (30 minutes - 2 hours after an anesthetic block, 2-3 months after neurotomy or botulinium toxin injection) allowing assessment of the responsiveness of the MSPMI. If the patient is not on these two situations, he will be included on the "simple evaluation group" and his participation will end.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity with respect to the Lance defintion (minimal score of 1 on the modified Ashworth scale)

Exclusion Criteria:

* Contraindication of ankle manipulation : fracture, phlebitis, bedsore
* amyotrophic lateral sclerosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Duration of the mobilization reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
range of motion (degree) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
maximal angular speed (degree.sec-1) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
torque peaque (N.m) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
work variability index (mJ.sec) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
area under the curve raw Work = f(time) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
area under the curve rectified Work = f(time) (J.sec) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
raw and averaged rectified EMG for Soleus and Gastrocnemius medialis (μV and μV.sec-1) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
Raw rectified EMG for Soleus (μv) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
Averaged rectified EMG for Gastrocnemius medialis (μv.sec-1) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
Averaged rectified EMG for Soleus (μv.sec-1) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
Maximal value of EMG for Gastrocnemius medialis (μv) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient
Maximal value of EMG for Soleus (μv) reproductibility coefficient | Day 0
  inter-rater intra-session reproductibility coefficient

SECONDARY OUTCOMES:
duration of the mobilization (sec) | Day0
  Patients of the 3 groups
duration of the mobilization (sec), | Day7
  Patients included in the "hospitalization group"
duration of the mobilization (sec), | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
duration of the mobilization (sec), | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
range of motion (degree), | Day0
  Patients of the 3 groups
range of motion (degree), | Day7
  Patients included in the "hospitalization group"
range of motion (degree), | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
range of motion (degree), | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
maximal angular speed (degree.sec-1) | Day 0
  Patients of the 3 groups
maximal angular speed (degree.sec-1) | Day 7
  Patients included in the "hospitalization group"
maximal angular speed (degree.sec-1) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
maximal angular speed (degree.sec-1) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
torque peaque (N.m) | Day 0
  Patients of the 3 groups
torque peaque (N.m) | Day 7
  Patients included in the "hospitalization group"
torque peaque (N.m) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
torque peaque (N.m) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
work variability index (mJ.sec) | Day0
  Patients of the 3 groups
work variability index (mJ.sec) | Day7
  Patients included in the "hospitalization group"
work variability index (mJ.sec) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
work variability index (mJ.sec) | 2 to 3 months after neurotomy or botulinium toxin injection
area under the curve raw Work = f(time) | Day 0
  Patients of the 3 groups
area under the curve raw Work = f(time) | Day 7
  Patients included in the "hospitalization group"
area under the curve raw Work = f(time) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
area under the curve raw Work = f(time) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
area under the curve rectified Work = f(time) (J.sec) | Day 0
  Patients of the 3 groups
area under the curve rectified Work = f(time) (J.sec) | Day 7
  Patients included in the "hospitalization group"
area under the curve rectified Work = f(time) (J.sec) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
area under the curve rectified Work = f(time) (J.sec) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
raw rectified EMG for Gastrocnemius medialis (μV and μV.sec-1) | Day 0
  Patients of the 3 groups
raw rectified EMG for Gastrocnemius medialis (μV and μV.sec-1) | Day 7
  Patients included in the "hospitalization group"
raw rectified EMG for Gastrocnemius medialis (μV and μV.sec-1) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
raw rectified EMG for Gastrocnemius medialis (μV and μV.sec-1) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
Averaged rectified EMG for Gastrocnemius medialis (μv.sec-1) | Day0
  Patients of the 3 groups
Averaged rectified EMG for Gastrocnemius medialis (μv.sec-1) | Day7
  Patients included in the "hospitalization group"
Averaged rectified EMG for Gastrocnemius medialis (μv.sec-1) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
Averaged rectified EMG for Gastrocnemius medialis (μv.sec-1) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
Raw rectified EMG for Soleus (μv) | Day 0
  Patients of the 3 groups
Raw rectified EMG for Soleus (μv) | Day 7
  Patients included in the "hospitalization group"
Raw rectified EMG for Soleus (μv) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
Raw rectified EMG for Soleus (μv) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
Averaged rectified EMG for Soleus (μv.sec-1) | Day 0
  Patients of the 3 groups
Averaged rectified EMG for Soleus (μv.sec-1) | Day 7
  Patients included in the "hospitalization group"
Averaged rectified EMG for Soleus (μv.sec-1) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
Averaged rectified EMG for Soleus (μv.sec-1) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
maximal value of EMG for Gastrocnemius medialis (μV) | Day0
  Patients of the 3 groups
maximal value of EMG for Gastrocnemius medialis (μV) | Day7
  Patients included in the "hospitalization group"
maximal value of EMG for Gastrocnemius medialis (μV) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
maximal value of EMG for Gastrocnemius medialis (μV) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
Maximal value of EMG for Soleus (μv) | Day 0
  Patients of the 3 groups
Maximal value of EMG for Soleus (μv) | Day 7
  Patients included in the "hospitalization group"
Maximal value of EMG for Soleus (μv) | 30minutes to 2 hours after an anesthesic block
  Patients included in the "treatment group" and treated by anesthesic block
Maximal value of EMG for Soleus (μv) | 2 to 3 months after neurotomy or botulinium toxin injection
  Patients included in the "treatment group" and treated by selective tibial neurotomy or toxin intramuscular injection
score on the modified Asworth scale | Day 0
  Patients of the 3 groups
modified Tardieu scale assigned by the evaluator | Day 0
  Patients of the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Perrouin-Verbe, PU-PH, Principal Investigator — Nantes CHU
Locations (1):
- Médecine Physique et Réadaptation Neurologique, Nantes, France

REFERENCES:
- [Background] Bar-On L, Aertbelien E, Molenaers G, Van Campenhout A, Vandendoorent B, Nieuwenhuys A, Jaspers E, Hunaerts C, Desloovere K. Instrumented assessment of the effect of Botulinum Toxin-A in the medial hamstrings in children with cerebral palsy. Gait Posture. 2014 Jan;39(1):17-22. doi: 10.1016/j.gaitpost.2013.05.018. Epub 2013 Jun 20. PMID 23791154
- [Background] Bar-On L, Van Campenhout A, Desloovere K, Aertbelien E, Huenaerts C, Vandendoorent B, Nieuwenhuys A, Molenaers G. Is an instrumented spasticity assessment an improvement over clinical spasticity scales in assessing and predicting the response to integrated botulinum toxin type a treatment in children with cerebral palsy? Arch Phys Med Rehabil. 2014 Mar;95(3):515-23. doi: 10.1016/j.apmr.2013.08.010. Epub 2013 Aug 27. PMID 23994052
- [Background] de Vlugt E, de Groot JH, Schenkeveld KE, Arendzen JH, van der Helm FC, Meskers CG. The relation between neuromechanical parameters and Ashworth score in stroke patients. J Neuroeng Rehabil. 2010 Jul 27;7:35. doi: 10.1186/1743-0003-7-35. PMID 20663189
- [Background] Schless SH, Desloovere K, Aertbelien E, Molenaers G, Huenaerts C, Bar-On L. The Intra- and Inter-Rater Reliability of an Instrumented Spasticity Assessment in Children with Cerebral Palsy. PLoS One. 2015 Jul 2;10(7):e0131011. doi: 10.1371/journal.pone.0131011. eCollection 2015. PMID 26134673
- [Background] Gaverth J, Sandgren M, Lindberg PG, Forssberg H, Eliasson AC. Test-retest and inter-rater reliability of a method to measure wrist and finger spasticity. J Rehabil Med. 2013 Jul;45(7):630-6. doi: 10.2340/16501977-1160. PMID 23695917
- [Background] Turk R, Notley SV, Pickering RM, Simpson DM, Wright PA, Burridge JH. Reliability and sensitivity of a wrist rig to measure motor control and spasticity in poststroke hemiplegia. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):684-96. doi: 10.1177/1545968308315599. Epub 2008 Sep 5. PMID 18776066